CLINICAL TRIAL: NCT03912220
Title: Evaluation of Nicotinamide Riboside in Prevention of Small Fiber Axon Degeneration and Promotion of Nerve Regeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Adelson Medical Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00210072
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Small Fiber Neuropathy
MeSH Terms: conditions — Small Fiber Neuropathy | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicotinamide Riboside (Experimental): Experimental group of participants will receive Nicotinamide riboside at a dose of 900 mg twice a day orally.
  Interventions: Drug: Nicotinamide riboside
- Placebo (Placebo Comparator): Study participants in the placebo arm will receive placebo pills that are similar in size and shape to the experimental group drug.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Nicotinamide riboside — The experimental arm will investigate the effects of nicotinamide riboside on nerve degeneration and regeneration.
  Arms: Nicotinamide Riboside
Drug: Placebo Oral Tablet — Placebo drug that looks like the experimental drug, nicotinamide riboside tablets.
  Arms: Placebo

SUMMARY:
This study will evaluate the effects of a nutritional supplement called nicotinamide riboside in preventing small fiber nerve degeneration that is experimentally induced by applying capsaicin to skin in otherwise healthy study participants. Furthermore, the effects on nerve regeneration will also be evaluated. The results will be compared to a placebo control drug.

DETAILED DESCRIPTION:
Small fiber neuropathy (SFN) is a type of peripheral neuropathy that affects the small unmyelinated fibers, including both somatic innervation of the skin and autonomic nerves. Although diabetes and prediabetes are the two most common causes, up to 50% of all SFN remain idiopathic. Currently there is no effective treatment that prevents it or reverses it through regeneration of nerve fibers.

Recent advances in understanding the molecular machinery that mediates Wallerian degeneration (i.e. degeneration of nerve fibers after physical transection) showed that key molecular players in this pathway and nicotinamide (NAD+) metabolites play a similar role in degeneration of axons in a distal-to-proximal manner seen in many peripheral neuropathies including SFN. Pre-clinical studies have shown that rapid depletion of NAD initiates a cascade of molecular events that leads to axon degeneration and that supplementation of a NAD precursor, nicotinamide riboside (NR) can prevent this degeneration.

In this study investigators plan to evaluate the ability of NR to prevent degeneration of small somatic sensory axons innervating the epidermis as well as its ability to promote regeneration of these same fibers in a human experimental model of nerve degeneration and regeneration. This experimental human model has been used previously to evaluate the rate of nerve degeneration and regeneration in several peripheral neuropathies and in healthy subjects.

Since NR is available as a nutritional supplement, if successful, this research can lead to development of a therapy for a variety of peripheral neuropathies very rapidly.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65
* BMI<32
* Normal neurological examination defined as Neuropathy Impairment Score <2

Exclusion Criteria:

* History of peripheral neuropathy
* Any peripheral neuropathy risk factor including diabetes, Vitamin B12 deficiency, HIV-infection, chronic kidney or hepatic disease, hypothyroidism, chemotherapy or other know neurotoxic exposure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Hoke, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicotinamide Riboside | Placebo
Started | 26 | 19
Completed | 26 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotinamide Riboside | Placebo | Total
Number analyzed (Participants) | 26 | 19 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 19 | 45
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 15 | 12 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 20 | 14 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 19 | 45
Baseline intraepidermal nerve fiber density [Median (Standard Deviation); unit: fibers/mm] | 10.75 (5) | 11.1 (3.9) | 10.9 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Denervation of Skin
Description: Examination of degree of loss of intraepidermal nerve fibers in the skin after experimental denervation by capsaicin. The skin biopsies will be stained for a pan-axonal marker and the number of intraepidermal nerve fibers per millimeter (mm) of skin will be counted and compared to baseline skin biopsy to determine the percent change in density of intraepidermal nerve fibers.
Time Frame: 2 days
Measure: Median (Full Range); unit: percent change
Arm/Group | Nicotinamide Riboside | Placebo
Number analyzed (Participants) | 26 | 19
percent change | 0.1 [0 to 0.8] | 0.1 [0 to 1.0]
Statistical Analysis 1: Comparison: Nicotinamide Riboside vs Placebo; Test type: Superiority; p = 0.33, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Reinnervation of Skin
Description: Examination of degree of re-innervation of skin after experimental denervation by capsaicin. The skin biopsies will be stained for a pan-axonal marker and the number of intraepidermal nerve fibers per mm of skin will be counted and compared to epidermal nerve fiber density after capsaicin application to determine the median density of intraepidermal nerve fibers.
Time Frame: 3 months
Measure: Median (Full Range); unit: intraepidermal nerve fibers per mm
Arm/Group | Nicotinamide Riboside | Placebo
Number analyzed (Participants) | 26 | 19
intraepidermal nerve fibers per mm | 7.4 [3 to 12.8] | 7.3 [3 to 11.8]
Statistical Analysis 1: Comparison: Nicotinamide Riboside vs Placebo; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Nicotinamide Riboside | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/19
Other Adverse Events (participants affected / at risk) | 0/26 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT03912220/Prot_SAP_000.pdf